CLINICAL TRIAL: NCT02807961
Title: Phase 1a, Randomized, Double-blinded, Placebo-controlled, Single-dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ELX-02 in Healthy Adult Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetics of ELX-02 in Healthy Adult Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Transferred study to Antwerp, Belgium
Sponsor: Eloxx Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EL-001
Record Dates: First submitted 2016-06-10; First posted 2016-06-21 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2017-08

CONDITIONS: Genetic Diseases; Nonsense Mutations
Keywords: Translational read through
MeSH Terms: conditions — Genetic Diseases, Inborn | interventions — ELX-02

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo comparator arm
  Interventions: Drug: Placebo
- Active treatment (Active Comparator): ELX-02, active comparator
  Interventions: Drug: ELX-02

INTERVENTIONS:
Drug: ELX-02 — Synthetic aminoglycoside
  Arms: Active treatment
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
This is the first study in humans of ELX-02, an advanced synthetic aminoglycoside optimized as a translational read-through drug (TRID) for the treatment of genetic conditions caused by nonsense. mutations. This is a classical Phase 1a study designed as a randomized, double-blinded, placebo-controlled, single dose escalation to evaluate the safety, tolerability and pharmacokinetics of ELX-02 in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following inclusion criteria to be eligible for enrollment in the study:

1. Be able and willing to provide written Informed Consent indicating that the subject has been informed of all pertinent aspects of the study.
2. Be willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Healthy female subjects and/or male subjects who, at the time of Screening, are between the ages of 18 and 45 years, inclusive.

   Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurements, 12-lead ECG and clinical laboratory tests.
4. Female subjects of non childbearing potential must meet at least one of the following criteria: Postmenopausal status, defined as: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; post-menopausal status will be confirmed by a serum FSH level, Have undergone a documented hysterectomy and/or bilateral oophorectomy, Have medically confirmed ovarian failure Female subjects of non-childbearing potential must agree to undergo pregnancy test at Screening.

   All other female subjects (including females with tubal ligations) will be considered to be of childbearing potential and may be enrolled if they have negative pregnancy tests on Screening and admission days and agree to use a reliable method of contraception for two weeks (14 days) before and four weeks (28 days) after dosing.

   Female subjects of childbearing potential must agree to undergo repeated pregnancy tests.

   Reliable methods of contraception include: Abstention from sexual intercourse, Established use of oral, inserted, injected, implanted or transdermal hormonal methods of contraception (provided the subject plans to remain on the same treatment throughout the entire study and has been using that hormonal contraceptive for an adequate period of time to ensure effectiveness), Copper-containing intrauterine device
5. Male subjects must be willing to use an effective method of contraception during the course of the study until 28 days after drug administration. These include condom, having undergone a vasectomy or abstain from sexual intercourse.
6. Be on no medications with potential to impair renal function, e.g., NSAIDs, or with ototoxic potential, e.g., quinine or salicylates.
7. Non-smoking and no use of any tobacco or nicotine products (by declaration) for a period of at least 6 months prior to Screening visit.
8. Normal renal function (MDRD GFR > 60 mL/min) based on serum creatinine concentration.
9. Negative HIV, HBsAg or HCV Ab serology tests at Screening.
10. No personal history of hearing loss, tinnitus, vertigo, imbalance and unsteadiness.
11. Normal Screening auditory and vestibular assessments.
12. Body Mass Index (BMI) of 19.0 to 30.0 Kg/m2.

Exclusion Criteria

Subjects with any of the following characteristics/conditions will not be included in the study:

1. Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or subjects who are the Sponsor employees directly involved in the conduct of the study.
2. Participation in another clinical trial within 6 months prior to dosing (calculated from the previous study's last doing day). If the previous trial involved agents with delayed effects or prolonged metabolism, a 12 months interval is required.
3. Evidence or history of clinically relevant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies,). This includes any acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or ELX-02 administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.
4. A positive urine drug screen (cannabinoids, amphetamines, benzodiazepines, and opiates), at Screening and on admission.
5. History of regular alcohol consumption (by declaration) exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 150 mL of wine or 360 mL of beer or 45 mL of hard liquor) within 6 months of Screening. A positive alcohol breath test on admission.
6. Screening supine blood pressure (BP) ≥ 140 mm Hg (systolic) or ≥ 90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP exceeds protocol-required limits, BP measurement should be repeated for up to two more times and the last BP value should be used to determine the subject's eligibility.
7. Screening supine 12-lead ECG demonstrating QTc >450 msec for men or >470 msec for women, or a QRS interval >120 msec.
8. Subjects with ANY abnormalities in clinical laboratory tests at Screening, considered by the Investigator as clinically relevant. In particular, subjects with ALT, AST and total bilirubin ≥ 1.5 upper limit of normal will be excluded.
9. Pregnant or breastfeeding female subjects.
10. Use of prescription or nonprescription drugs, vitamins, herbal and/or dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to administration of ELX-02. As an exception, acetaminophen/paracetamol may be used at doses of ≤ 2 g/day. Aspirin and NSAIDS should not be administered within 1 week of study dose. Limited use of non-prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the Sponsor.
11. Subjects who donated blood or received blood or plasma derivatives in the 3 months preceding study drug administration.
12. Known allergy or hypersensitivity to any drug and/or to any of the excipients of ELX-02.
13. Subjects with an inability to communicate well with the Investigators and CRC staff (e.g., language problem, poor mental development).
14. Subjects with any acute medical situation (e.g. acute infection) within 48 hours prior to Day 1, which is considered of significance by the Principal Investigator.
15. Subjects with any history of ear disease or surgeries, dizziness or ongoing tinnitus.
16. Subjects with any abnormality on physical examination by an ENT specialist at screening that indicates the presence of a vestibular pathology, conductive hearing loss or balance problem.
17. Subjects with audiometry results as follows: any pure-tone threshold >25dB, inter-ear difference in any frequency of ≥ 20dB, word recognition score (discrimination) <92%.
18. Abnormal ENG/VNG [as indicated by a cumulative response of <12 degrees to caloric testing (response to warm and cold stimulation united) in either ear] or abnormal c/v HIT.
19. DHI-H score >16
20. THI-H score >14

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 0-10 days
  Incidence and characteristics of adverse events occurring following single doses of ELX-02
Pharmacokinetics | 0-10 days
  The following PK parameters will be calculated based on ELX-02 plasma concentrations: Cmax, Tmax, AUC24h, AUCinf, AUC144h, t½, mean residence time (MRT), volume of distribution (Vd), clearance (CL), absolute bioavailability (F) and an estimation of ELX-02 dose linearity of PK parameters. The following parameters will be calculated based on ELX-02 urine concentrations: urinary mass excretion of ELX-02 (in mass and %dose) and cumulated urinary excretion (in % dose) for each collection interval and total renal clearance. The following parameters will be calculated from the individual urine drug concentrations: Ae, Ae0-12h, Ae12-24h, Ae24-48h, Ae0-48h, fe.